CLINICAL TRIAL: NCT04526119
Title: Z-338 Phase III Trial - Evaluation of Pharmacokinetics, Efficacy and Safety in Paediatric Patients With Functional Dyspepsia
Brief Title: A Phase III Trial of Z-338 in Paediatric Patients With Functional Dyspepsia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z-338-07
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Z-338 (Experimental)
  Interventions: Drug: Acotiamide hydrochloride hydrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acotiamide hydrochloride hydrate — A white film-coated tablet containing 100 mg Z-338 Administered orally, one tablet a time and three times a day before meals for 28 days in the double-blind phase Administered orally, one tablet a time and three times a day before meals for 28 days in the open-label phase
  Arms: Z-338
Drug: Placebo — A white film-coated tablet not containing 100 mg Z-338 Administered orally, one tablet a time and three times a day before meals for 28 days in the double-blind phase
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics, efficacy and safety of Z-338 of pediatric patients with functional dyspepsia (FD).

In Part 1, the pharmacokinetics and safety of single oral dose of Z-338 100 mg are evaluated.

In Part 2, the efficacy and safety of Z-338 100 mg orally 3 times daily before meals are evaluated.

Part 2 is comprised by the double-blind phase and the open-label phase. In the double-blind phase, subjects will take Z-338 or placebo for 28 days. In the open-label phase, all subjects will take Z-338 for 28 days.

ELIGIBILITY:
Main Inclusion Criteria:

Part 1& Part 2

* Subjects aged from nine to 17 years (from nine to 14 years in Part 1), on the day the informed consent is signed.
* Subjects with a diagnosis of FD as defined by the Rome IV Criteria.
* Subjects who have postprandial fullness, upper abdominal bloating or early satiation.

Part 2 only

* Subjects who have postprandial fullness, upper abdominal bloating or early satiation during with a certain severity during a week prior to the day of randomization.

Main Exclusion Criteria:

Part 1&Part 2

* Subject who have organic diseases of the gastrointestinal tract or gastrointestinal bleeding within 24 weeks prior to informed consent.
* Subject who have received Helicobacter pylori eradication therapy within 24 weeks prior to informed consent, or subjects who is defined as Helicobacter pylori-positive within 4 weeks prior to or on the day the informed consent is signed.
* Subjects who have alarm symptom on the day the informed consent is signed.
* Subjects who have food allergy of unknown origin or uncontrolled food allergy.

Part 2 only

* Subject taking drugs used for FD within 2 weeks prior to the day of randomization (excluding proton pump inhibitors)
* Subject taking proton pump inhibitors within 4 weeks prior to the day of randomization.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cmax of single dose Z-338 before meal | The 1 day of single dose
AUC up to 8 hours after administration of single dose Z-338 before meal | The 1 day of single dose
Elimination rate of three symptoms (Postprandial fullness, Upper abdominal bloating and Early satiation) | At week 4 of treatment or treatment discontinuation
Overall responder rate by the Overall Treatment Evaluation (OTE) scale | At week 4 of treatment or treatment discontinuation

SECONDARY OUTCOMES:
Elimination rate of each symptom | Weekly from the day of randomization to Week 8
Average severity score of each symptom | Weekly from the day of randomization to Week 8
Worst severity score of each symptom | Weekly from the day of randomization to Week 8
Weekly responder rate by the OTE scale | Weekly from the day of randomization to Week 8
Incidence of adverse events | 8-weeks study period
Incidence of adverse drug reactions | 8-weeks study period

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Shibasaki, Study Director — Zeria Pharmaceutical
Locations (1):
- Zeria Investigative Site, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No